CLINICAL TRIAL: NCT00898950
Title: The Links Between Dysglycaemia, Insulin Resistance, Endothelial Function, Inflammation and Oxidative Stress: Effect of Different Doses of Aspirin in Subjects With Type-2 Diabetes and High Cardiovascular Risk
Brief Title: Effects of Different Doses of Aspirin on Pathophysiological Markers in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Portsmouth (Other)
Responsible Party: Dr MH Cummings, Portsmouth Hospitals NHS Trust & University of Portsmouth
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2004-001418-14
Record Dates: First submitted 2009-05-11; First posted 2009-05-12 (Estimated); Last update posted 2009-05-12 (Estimated); Status verified 2009-05

CONDITIONS: Diabetes Type 2
Keywords: diabetes; aspirin; oxidative stress; insulin resistance; endothelial function; inflammation; photoplethysmography; dysglycaemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance; Inflammation | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Aspirin low dose (Experimental): Effects of using aspirin 75 mgs/day for 2 weeks.
  Interventions: Drug: Aspirin
- Aspirin medium dose (Experimental): Effects of using aspirin 300 mgs/day
  Interventions: Drug: Aspirin
- aspirin high dose (Experimental): aspirin 900mgs QID orally for 2 weeks
  Interventions: Drug: Aspirin
- placebo (Placebo Comparator)
  Interventions: Other: placebo tablet

INTERVENTIONS:
Drug: Aspirin — Aspirin 75mgs/day orally for 2 weeks.
  Other Names: acetyl salicylic acid
  Arms: Aspirin low dose
Drug: Aspirin — 300mgs/day orally for 2 weeks
  Other Names: acetyl salicylic acid
  Arms: Aspirin medium dose
Drug: Aspirin — aspirin 900mgs QID orally for 2 weeks
  Other Names: acetyl salicylic acid
  Arms: aspirin high dose
Other: placebo tablet — placebo tablet with lactose and excipients.
  Arms: placebo

SUMMARY:
This study was set up to assess the effects of different doses of aspirin when compared with placebo (dummy drug), used sequentially over a 2 week study period with a 2 week wash-out (rest period) in between, in people with type-2 diabetes and high cardiovascular risk. Specifically, its effects on different factors which are thought to contribute to diabetes such as insulin resistance (body's ability to effectively use insulin), dysglycaemia (excess glucose in the blood), oxidative stress (effects from accumulation of by-products of metabolism), endothelial function (function of lining of blood vessels) and inflammation were studied.

ELIGIBILITY:
Inclusion Criteria:

* diabetes type 2
* age > 18 and < 70
* high cardiovascular risk

Exclusion Criteria:

* presence of active/established cardiovascular disease (ischaemic heart disease, cerebrovascular disease or peripheral vascular disease)
* insulin treatment
* patients with known peptic ulcer disease or those on anti-coagulation
* significant renal impairment
* aspirin intolerance
* use of anticoagulants
* significant liver disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2004-08; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Change in markers of oxidative stress, endothelial function, glycaemic control, and insulin resistance | 2 weeks

SECONDARY OUTCOMES:
Change in inflammatory markers | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rajeev P Raghavan, MBBS, MRCP, Principal Investigator — Portsmouth Hospitals NHS Trust; Michael H Cummings, MD, FRCP, Study Director — Portsmouth Hospitals NHS TRust & University of Portsmouth
Locations (2):
- United Kingdom (2):
  - School of Pharmacy and Biomedical Sciences, University of Posrtmouth, Portsmouth, Hampshire
  - Diabetes Centre, Queen Alexandra Hospital, Portsmouth Hospitals NHS Trust, Portsmouth, Hampshire

REFERENCES:
- [Derived] Raghavan RP, Laight DW, Cummings MH. Aspirin in type 2 diabetes, a randomised controlled study: effect of different doses on inflammation, oxidative stress, insulin resistance and endothelial function. Int J Clin Pract. 2014 Feb;68(2):271-7. doi: 10.1111/ijcp.12310. Epub 2013 Dec 22. PMID 24372992